CLINICAL TRIAL: NCT04728893
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of MK-1026 in Participants With Hematologic Malignancies
Brief Title: Efficacy and Safety of Nemtabrutinib (MK-1026) in Participants With Hematologic Malignancies (MK-1026-003)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026-003; MK-1026-003 (Other: MSD); 2023-504931-42-00 (Registry Identifier: EU CT); U1111-1290-4004 (Registry Identifier: UTN); 2020-002324-36 (EudraCT Number)
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hematologic Malignancies; Waldenstroms Macroglobulinaemia; Non-Hodgkins Lymphoma; Chronic Lymphocytic Leukaemia
MeSH Terms: conditions — Hematologic Neoplasms; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin; Leukemia, B-Cell | interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nemtabrutinib (Experimental): Participants receive nemtabrutinib orally once daily (QD) until progressive disease (PD) or discontinuation.
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Nemtabrutinib tablets administered orally QD.
  Other Names: ARQ 531; MK-1026

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nemtabrutinib (formerly ARQ 531) in participants with hematologic malignancies of chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL), Richter's transformation, marginal zone lymphoma (MZL), mantle cell lymphoma (MCL), follicular lymphoma (FL), and Waldenström's macroglobulinemia (WM).

DETAILED DESCRIPTION:
This study will be performed in 2 parts: Dose Escalation and Confirmation (Part 1) and Cohort Expansion (Part 2). Following determination of the recommended phase 2 dose (RP2D) in Part 1, the study plans to proceed with Part 2 using 8 disease-specific expansion cohorts (Cohorts A to H).

ELIGIBILITY:
Inclusion Criteria:

* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 within 7 days before C1D1 (the first dose of study treatment)
* Has a life expectancy of at least 3 months, based on the investigator assessment
* Has the ability to swallow and retain oral medication
* Participants who are Hepatitis B surface antigen (HBsAg)-positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization
* Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening
* Has adequate organ function
* Male participants agree to refrain from donating sperm and agree to either remain abstinent from penile-vaginal intercourse as their preferred and usual lifestyle OR agree to use contraception, during the intervention period and for at least the time required to eliminate the study intervention after last dose of study intervention
* Female participants assigned female sex at birth who are not pregnant or breastfeeding are eligible to participate if not a participant of childbearing potential (POCBP), or if a POCBP they either use a contraceptive method that is highly effective OR remain abstinent from penile-vaginal intercourse as their preferred and usual lifestyle during the intervention period and for at least to eliminate study intervention after the last dose of study intervention
* Participants with Human immunodeficiency virus (HIV) are eligible if they meet all of the following: the CD4 count is >350 cells/uL at screening, the HIV viral load is below the detectable level, are on a stable ART regimen for at least 4 weeks prior to study entry, and are compliant with their ART

Part 1 and Part 2 (Cohorts A to C and J)

* Has a confirmed diagnosis of Chronic lymphocytic leukemia/ Small lymphocytic lymphoma (CLL/SLL) with

  * At least 2 lines of prior therapy (Part 1 only)
  * Part 2 Cohort A: CLL/SLL participants who are relapsed or refractory to prior therapy with a covalent, irreversible Bruton's tyrosine kinase inhibitor (BTKi), and a B-cell lymphoma 2 inhibitor (BCL2i). CLL participants must have received and failed, been intolerant to, or determined by their treating physician to be a poor phosphoinositide 3-kinase inhibitor (PI3Ki) candidate or ineligible for a PI3Ki per local guidelines
  * Part 2 Cohort B: CLL/SLL participants who are relapsed or refractory following at least 1 line of prior therapy and are BTKi treatment naive
  * Part 2 Cohort C: CLL/SLL participants with 17p deletion or tumor protein p53 (TP53) mutation who are relapsed or refractory following at least 1 line of prior therapy
  * Part 2 Cohort J: CLL/SLL participants whose disease relapsed or was refractory to prior therapy with a covalent/irreversible BTKi and BCL2i. NOTE: As of Protocol Amendment 09, at least 10 CLL/SLL participants whose disease relapsed or was refractory to prior therapy with a covalent/irreversible BTKi, BCL2i and noncovalent/reversible BTKi (all three classes of therapies are required) will be enrolled into Cohort J
  * Has active disease for CLL/SLL clearly documented to initiate therapy
  * For SLL participants in Part 2: Has evaluable core or excisional lymph node biopsy for biomarker analysis from an archival or newly obtained biopsy or bone marrow aspirate at Screening (optional for participants enrolling in Part 1)

Part 2 (Cohorts D to G)

- Has a confirmed diagnosis of and meets the following prior therapy requirements:

* Participants with Richter's transformation who are relapsed or refractory following at least 1 line of prior therapy (Cohort D)
* Participants with pathologically confirmed Mantle-cell lymphoma (MCL), documented by either overexpression of cyclin D1 or t (11;14), who are relapsed or are refractory to chemoimmunotherapy and a covalent irreversible BTKi (Cohort E)
* Participants with Marginal zone lymphoma (MZL) (including splenic, nodal, and extra nodal MZL) who are relapsed or refractory to at least one prior line of systemic therapy including an anti-CD20-based regimen
* Participants with Follicular lymphoma (FL) who are relapsed or refractory to chemoimmunotherapy and immunomodulatory agents (such as lenalidomide based regimen) (Cohort G)
* Have measurable disease defined as at least 1 lesion that can be accurately measured in at least 2 dimensions with spiral Computed tomography (CT) scan
* Has a lymph node biopsy for biomarker analysis from an archival or newly obtained biopsy or bone marrow aspirate (Cohort D) at Screening

Part 2 (Cohort H): confirmed diagnosis of Waldenström's macroglobulinemia (WM); participants who are relapsed or refractory to standard therapies for WM including chemoimmunotherapy and a covalent irreversible BTKi

* Has active disease defined as 1 of the following: systemic symptoms, physical findings, laboratory abnormalities, coexisting disease
* Has measurable disease, satisfying any of the following: at least 1 lesion that can be accurately measured in at least 2 dimensions with spiral CT scan (minimum measurement must be >15 mm in the longest diameter or >10 mm in the short axis); IgM ≥450 mg/dL; or bone marrow infiltration of 10%
* Has fresh bone marrow aspirate or a lymph node biopsy for biomarker analysis at Screening or a lymph node biopsy from an archival

Exclusion Criteria:

* Has active HBV/HCV infection (Part 1 and Part 2)
* Has a history of malignancy ≤3 years before providing documented informed consent. Participants with basal cell carcinoma of skin, squamous cell carcinoma of skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potential curative therapy are not excluded. Participants with low-risk, early-stage prostate cancer (T1-T2a, Gleason score ≤6, and prostate-specific antigen <10 ng/mL) either treated with definitive intent or untreated in active surveillance with SD are not excluded
* Has active central nervous system (CNS) disease
* Has an active infection requiring systemic therapy
* Has received prior systemic anti-cancer therapy within 5 half-lives or 4 weeks (if prior therapy was a monoclonal antibody) before C1D1
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has any clinically significant gastrointestinal abnormalities that might alter absorption
* History of severe bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-04-05 (Actual); Primary Completion 2029-01-04 (Estimated); Study Completion 2029-01-04 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants experiencing dose-limiting toxicities (DLTs) | Up to ~56 days (Cycles 1-2, cycle = 28 days)
  DLTs will be defined as toxicities observed during the first 2 cycles (8 weeks) of Part 1 and include: Grade ≥3 nonhematologic toxicity (except Grade 3 nausea, vomiting, diarrhea, rash, fatigue, and uncontrolled hypertension which will not be considered a DLT unless lasting ≥72 hours despite optimal supportive care); Grade 4 hematologic toxicity lasting >7 days (except Grade 3 lymphocytosis, Grade 4 platelet count decreased of any duration, or Grade 3 platelet count decreased if associated with bleeding); any Grade 3 or Grade 4 nonhematologic laboratory abnormality if values result in drug-induced liver injury, or medical intervention is required, or the abnormality leads to hospitalization, or the abnormality persists for >1 week (with exceptions); missing >25% of nemtabrutinib doses as a result of drug-related adverse events (AEs) during the first 2 cycles (8 weeks); Grade 5 toxicity.
Part 1: Number of participants experiencing adverse events (AEs) | Up to ~71 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing AEs will be reported for Part 1.
Part 1: Number of participants discontinuing study treatment due to AEs | Up to ~42 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study treatment due to an AE will be reported for Part 1.
Part 2: Objective Response Rate (ORR) per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria 2018 as assessed by independent central review (ICR) | Up to ~61 months
  ORR per iwCLL 2018 criteria is defined as the percentage of participants achieving a complete response (CR), complete response with incomplete bone marrow recovery (CRi), nodular partial response (nPR), or partial response (PR). CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Part 2: ORR per Lugano criteria 2014 as assessed by ICR | Up to ~61 months
  ORR per Lugano criteria 2014 is defined as the percentage of participants achieving a CR or PR. CR defined as EITHER CR by imaging (computed tomography [CT]): all lymph nodes normal (none ≥15 mm) and normal liver and spleen OR complete metabolic response (CMR): score of 1, 2 or 3 on the 5-point scale assessing fluorodeoxyglucose (FDG) metabolic activity in lymphomatous lesions (ranging from 1=no uptake above background to 5=uptake markedly higher than liver) AND bone marrow (BM) normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in the sum of the product of diameters [SPD] of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR Partial Metabolic Response (PMR) with score of 4 or 5 on the FDG 5-point scale (with no new lesions) and decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.
Part 2: ORR per International Workshop on Waldenström's Macroglobulinemia (IWWM) criteria 2014 as assessed by ICR | Up to ~71 months
  ORR per IWWM criteria 2014 is defined as the percentage of participants achieving a CR, very good partial response (VGPR), or PR. CR is defined as all lymph nodes are normal in size (none ≥15 mm), liver and spleen normal in size, serum immunoglobulin M (IgM) values in the normal range, disappearance of monoclonal protein by immunofixation (confirmation needed with a second immunofixation at any subsequent timepoint), and no histological evidence of BM involvement. VGPR is defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline), ≥50% decrease from baseline in the abnormal portion of the spleen (if previously abnormal), and ≥90% decrease from baseline in serum IgM, or serum IgM values in normal range. PR is defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline), ≥50% decrease from baseline in serum IgM, and ≥50% decrease from baseline in the abnormal portion of the spleen (if previously abnormal).

SECONDARY OUTCOMES:
Part 1: Area Under the Curve (AUC) of Nemtabrutinib | At designated time points (up to ~57 days)
  Blood samples will be obtained at designated time points during Part 1 for the assessment of nemtabrutinib AUC (Day 1 of Cycles 1 and 2: Pre-dose, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2, 4, and 6 hours post-dose [up to ~57 days]). Each cycle is 28 days.
Part 1: Minimum Concentration (Cmin) of Nemtabrutinib | At designated time points (up to ~57 days)
  Blood samples will be obtained at designated time points during Part 1 for the assessment of nemtabrutinib Cmin (Day 1 of Cycles 1 and 2: Pre-dose, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2, 4, and 6 hours post-dose [up to ~57 days]). Each cycle is 28 days.
Part 1: Maximum Concentration (Cmax) of Nemtabrutinib | At designated time points (up to ~57 days)
  Blood samples will be obtained at designated time points during Part 1 for the assessment of nemtabrutinib Cmax (Day 1 of Cycles 1 and 2: Pre-dose, 2, 4, 6, 8, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2, 4, and 6 hours post-dose [up to ~57 days]). Each cycle is 28 days.
Part 1: ORR per iwCLL criteria 2018 as assessed by ICR | Up to ~71 months
  ORR per iwCLL 2018 criteria is defined as the percentage of participants achieving a CR, CRi, nPR, or PR. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Part 1: Duration of Response (DOR) per iwCLL criteria 2018 as assessed by ICR | Up to ~71 months
  For participants with CR, CRi, nPR, or PR per iwCLL 2018 criteria, DOR is defined as the time from the first documented evidence of objective response until PD or death due to any cause, whichever occurs first. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Part 2: Number of participants experiencing AEs | Up to ~61 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing AEs will be reported for Part 2.
Part 2: Number of participants discontinuing study treatment due to AEs | Up to ~42 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants discontinuing study treatment due to an AE will be reported for Part 2.
Part 2: AUC of Nemtabrutinib | At designated time points (up to ~57 days)
  Blood samples will be obtained at designated time points during Part 2 for the assessment of nemtabrutinib AUC (Day 1 of Cycles 1, 2, and 3: Pre-dose, 2, 4, 6, hours post-dose [up to ~57 days]). Each cycle is 28 days.
Part 2: Cmin of Nemtabrutinib | At designated time points (up to ~57 days)
  Blood samples will be obtained at designated time points during Part 2 for the assessment of nemtabrutinib Cmin (Day 1 of Cycles 1, 2, and 3: Pre-dose, 2, 4, 6, hours post-dose [up to ~57 days]). Each cycle is 28 days.
Part 2: Cmax of Nemtabrutinib | At designated time points (up to ~57 days)
  Blood samples will be obtained at designated time points during Part 2 for the assessment of nemtabrutinib Cmax (Day 1 of Cycles 1, 2, and 3: Pre-dose, 2, 4, 6, hours post-dose [up to ~57 days]). Each cycle is 28 days.
Part 2: DOR per iwCLL criteria 2018 as assessed by ICR | Up to ~61 months
  For participants with CR, CRi, nPR, or PR per iwCLL 2018 criteria, DOR is defined as the time from the first documented evidence of objective response until disease progression or death due to any cause, whichever occurs first. CR is defined as meeting the following criteria: no lymph nodes >1.5 cm, spleen size <13 cm, liver normal; no constitutional symptoms, normal lymphocyte count, platelets ≥100 x 10^9/L; hemoglobin ≥11 g/dL; and normocellular marrow (no CLL cells or B lymphoid nodules). CRi is defined as meeting CR criteria but with hypocellular bone marrow. nPR is defined as having features of CR but with lymphoid nodules in the marrow. PR is defined as ≥50% decrease in ≥2 of the following: lymph nodes, liver and/or spleen size, lymphocytes PLUS ≥1 of the following met: platelets ≥100 x 10^9/L or ≥50% increase from screening, hemoglobin >11 g/dL or ≥50% increase from screening, CLL cells or B lymphoid nodules in marrow.
Part 2: DOR per Lugano criteria 2014 as assessed by ICR | Up to ~61 months
  For participants with CR or PR per Lugano criteria 2014, DOR is defined as the time from the first documented evidence of objective response until PD or death due to any cause, whichever occurs first. CR defined as EITHER CR by imaging (CT): all lymph nodes normal (none ≥15 mm) and normal liver and spleen OR CMR: score of 1, 2 or 3 on the 5-point scale assessing FDG metabolic activity in lymphomatous lesions (ranging from 1=no uptake above background to 5=uptake markedly higher than liver and/or new lesions) AND BM normal by morphology. PR defined as EITHER PR by imaging (CT) with ≥50% decrease in the SPD of target lesions, no worsening of nontarget lesions, no new lesions and ≥50% spleen abnormal portion OR PMR with score of 4 or 5 on the FDG 5-point scale (with no new lesions) and decreased overall uptake AND residual BM abnormalities; OR CR by imaging with residual BM abnormalities; OR PR by imaging without residual BM abnormalities.
Part 2: DOR per IWWM criteria 2014 as assessed by ICR | Up to ~61 months
  For participants with CR, VGPR, or PR per IWWM criteria 2014, DOR defined as the time from first documented evidence of objective response until PD or death due to any cause, whichever occurs first. CR defined as all lymph nodes normal in size (none ≥15 mm), liver and spleen normal in size, serum IgM values in normal range, disappearance of monoclonal protein by immunofixation (confirmation needed with second immunofixation at any subsequent timepoint), and no histological evidence of BM involvement. VGPR defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline), ≥50% decrease from baseline in abnormal portion of the spleen (if previously abnormal), and ≥90% decrease from baseline in serum IgM, or serum IgM values in normal range. PR is defined as ≥50% decrease from baseline in SPD of lymph nodes (if abnormal at baseline), ≥50% decrease from baseline in serum IgM, and ≥50% decrease from baseline in abnormal portion of the spleen (if previously abnormal).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (121):
- United States (11):
  - Highlands Oncology Group ( Site 2728), Springdale, Arkansas
  - University of California San Diego Moores Cancer Center ( Site 2717), La Jolla, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA-Hematology and Medical Oncology ( Site 2724), Torrance, California
  - Colorado Blood Cancer Institute ( Site 2726), Denver, Colorado
  - The University of Louisville, James Graham Brown Cancer Center ( Site 2729), Louisville, Kentucky
  - Mayo Clinic - Rochester ( Site 2706), Rochester, Minnesota
  - Astera Cancer Care ( Site 2732), East Brunswick, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 2704), Hackensack, New Jersey
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 2708), Fargo, North Dakota
  - UT Southwestern-Harold C. Simmons Cancer Center ( Site 2730), Dallas, Texas
  - Medical Oncology Associates (Summit Cancer Centers) ( Site 2710), Spokane, Washington
- Argentina (6):
  - Hospital Aleman ( Site 0102), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC) ( Site 0103), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos ( Site 0112), Rosario, Santa Fe Province
  - FUNDALEU ( Site 0104), Caba
  - Hospital Privado Universitario de Córdoba ( Site 0107), Córdoba
  - Fundacion Centro Oncologico de Integración Regional-Medical Oncology ( Site 0110), Mendoza
- Australia (3):
  - Nepean Hospital-Nepean Cancer Care Centre ( Site 0204), Sydney, New South Wales
  - Box Hill Hospital ( Site 0203), Box Hill, Victoria
  - Sir Charles Gairdner Hospital ( Site 0200), Nedlands, Western Australia
- Brazil (4):
  - Hospital das Clinicas FMUSP-Pesquisa Clínica Hematologia ( Site 0303), São Paulo, São Paulo
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0300), Rio de Janeiro
  - BP - A Beneficencia Portuguesa de São Paulo ( Site 0302), São Paulo
  - Hospital Paulistano - Amil Clinical Research ( Site 0311), São Paulo
- Canada (5):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 0401), Calgary, Alberta
  - The Ottawa Hospital ( Site 0404), Ottawa, Ontario
  - Princess Margaret Cancer Centre-Division of Medical Oncology and Hematology ( Site 0406), Toronto, Ontario
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0403), Montreal, Quebec
  - Jewish General Hospital ( Site 0400), Montreal, Quebec
- China (19):
  - Anhui Provincial Hospital ( Site 2808), Hefei, Anhui
  - Peking University Third Hospital-Hematology ( Site 2827), Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University ( Site 2825), Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center-Internal Medicine ( Site 2824), Guangzhou, Guangdong
  - Guangxi Medical University - Liuzhou Renmin Hospital ( Site 2817), Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 2814), Nanning, Guangxi
  - Henan Cancer Hospital-hematology department ( Site 2802), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 2816), Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University ( Site 2820), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 2822), Changsha, Hunan
  - Jiangsu Province Hospital ( Site 2823), Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 2818), Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 2815), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 2803), Changchun, Jilin
  - Fudan University Shanghai Cancer Center ( Site 2801), Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University ( Site 2821), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University ( Site 2810), Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Unio ( Site 2800), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 2826), Hangzhou, Zhejiang
- Czechia (2):
  - Fakultní nemocnice Brno Bohunice-Interni hematologicka a onkologicka klinika ( Site 0600), Brno, Brno-mesto
  - Fakultni nemocnice Hradec Kralove ( Site 0601), Hradec Králové
- Denmark (4):
  - Aarhus University Hospital ( Site 0702), Aarhus N, Central Jutland
  - Aalborg Universitetshospital ( Site 0703), Aalborg, North Denmark
  - Sjaellands Universitetshospital Roskilde ( Site 0701), Roskilde, Region Sjælland
  - Odense University Hospital ( Site 0705), Odense C, Region Syddanmark
- France (5):
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet ( Site 0810), Nice, Alpes-Maritimes
  - Centre Hospitalier Lyon-Sud ( Site 0804), Pierre-Bénite, Auvergne-Rhône-Alpes
  - Institut Paoli-Calmettes ( Site 0803), Marseille, Bouches-du-Rhone
  - Centre Hospitalier de Versailles ( Site 0809), Le Chesnay, Yvelines
  - Hopital Saint Louis ( Site 0805), Paris
- Germany (4):
  - Universitaetsklinikum Ulm. ( Site 0906), Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Koeln ( Site 0901), Cologne, North Rhine-Westphalia
  - St. Marien-Krankenhaus Siegen ( Site 0914), Siegen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus ( Site 0902), Dresden, Saxony
- Hungary (4):
  - Pecsi Tudomanyegyetem Altalanos Orvostudomanyi Kar ( Site 1202), Pécs, Baranya
  - Debreceni Egyetem Klinikai Kozpont ( Site 1201), Debrecen, Hajdú-Bihar
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház ( Site 1206), Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Orszagos Onkologiai Intezet ( Site 1200), Budapest
- Ireland (2):
  - Beaumont Hospital ( Site 2900), Dublin
  - University Hospital Limerick ( Site 2903), Limerick
- Israel (7):
  - Ha Emek Medical Center ( Site 1305), Afula
  - Soroka Medical Center ( Site 1307), Beersheba
  - Rambam Medical Center ( Site 1301), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 1300), Jerusalem
  - Chaim Sheba Medical Center ( Site 1302), Ramat Gan
  - Kaplan Medical Center ( Site 1304), Rehovot
  - Sourasky Medical Center ( Site 1303), Tel Aviv
- Italy (8):
  - Istituto Tumori Giovanni Paolo II ( Site 1409), Bari
  - A.O. Universitaria Policlinico S. Orsola-Malpighi ( Site 1400), Bologna
  - ASST Spedali Civili di Brescia ( Site 1408), Brescia
  - IRCCS Ospedale San Raffaele ( Site 1402), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 1403), Napoli
  - Fondazione IRCCS Policlinico San Matteo ( Site 1407), Pavia
  - IRCCS - Arcispedale Santa Maria Nuova ( Site 1405), Reggio Emilia
  - Policlinico Umberto I ( Site 1404), Roma
- Poland (5):
  - Pratia MCM Krakow ( Site 1601), Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny-Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku ( Site 1606), Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Kilinka Onkologii I Hematologii ( Site 1608), Warsaw, Masovian Voivodeship
  - Szpital Wojewódzki w Opolu-Hematology Department ( Site 1607), Opole, Opole Voivodeship
  - Szpitale Pomorskie Sp. z o.o. ( Site 1600), Gdynia, Pomeranian Voivodeship
- Romania (4):
  - Spitalul Clinic Colțea ( Site 1805), Bucharest, București
  - Ovidius Clinical Hospital ( Site 1804), Ovidiu, Constanța County
  - Centrul de Diagnostic si Tratament Oncologic Brasov ( Site 1802), Brasov
  - Institutul Regional de Oncologie Iasi ( Site 1801), Iași
- South Korea (2):
  - Severance Hospital Yonsei University Health System ( Site 2201), Seoul
  - Samsung Medical Center ( Site 2200), Seoul
- Spain (7):
  - Instituto Catalan de Oncologia ICO - Hospital Duran i Reynals ( Site 2000), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Salamanca ( Site 2002), Salamanca, Castille and León
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 2005), A Coruña, La Coruna
  - Hospital General Universitario de Alicante ( Site 2007), Alicante
  - Hospital Universitari Vall d'Hebron ( Site 2001), Barcelona
  - Hospital Universitario 12 de Octubre ( Site 2003), Madrid
  - Hospital Puerta de Hierro ( Site 2009), Madrid
- Switzerland (2):
  - Inselspital Bern ( Site 2303), Bern, Canton of Bern
  - Istituto Oncologica della Svizzera Italiana (IOSI) ( Site 2302), Bellinzona, Canton Ticino
- Turkey (Türkiye) (5):
  - Mega Medipol-Hematology ( Site 2406), Stanbul, Istanbul
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi ( Site 2400), Ankara
  - VKV Amerikan Hastanesi ( Site 2403), Istanbul
  - Sisli Florence Nightingale Hastanesi ( Site 2407), Istanbul
  - Dokuz Eylül Üniversitesi-Hematology ( Site 2402), Izmir
- Ukraine (4):
  - MNPE ClinCenter of Oncology,Hematology,Transplantology and Palliative Care of CherkasyRegCouncil ( Site 2509), Cherkassy, Cherkasy Oblast
  - Communal non-profit enterprise "Regional clinical hospital o-Hematology Department ( Site 2510), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Instit. of Blood Transfusion Medicine of the National Academy ( Site 2506), Lviv, Lviv Oblast
  - National Cancer Institute ( Site 2507), Kyiv
- United Kingdom (8):
  - Bristol Haematology and Oncology Centre ( Site 2610), Bristol, Bristol, City of
  - Nottingham University Hospitals NHS Trust. City Hospital Campus ( Site 2601), Nottingham, England
  - GenesisCare - Windsor ( Site 2608), Windsor, England
  - Sarah Cannon Research Institute UK ( Site 2612), London, London, City of
  - GenesisCare - Oxford ( Site 2607), Oxford, Oxfordshire
  - GenesisCare - Cambridge ( Site 2611), Newmarket, Suffolk
  - The Royal Marsden NHS Foundation Trust. ( Site 2606), Sutton, Surrey
  - The Christie NHS Foundation Trust ( Site 2602), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26308&tenant=MT_MSD_9011